CLINICAL TRIAL: NCT02534142
Title: Colonoscopy Followup After Positive Fecal Occult Blood Test- Understanding Barriers to Adherence
Status: Completed | Type: Observational
Sponsor: Meuhedet. Healthcare Organization (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 01-20-05-15
Record Dates: First submitted 2015-07-28; First posted 2015-08-27 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Completed followup: All members aged 50-74 who completed a fecal occult blood test between 1/1/2014 and 1/1/2015, who had a positive result and had a colonoscopy following the result.
- Did not complete followup: All members aged 50-74 who completed a fecal occult blood test between 1/1/2014 and 1/1/2015, who had a positive result and did not have a colonoscopy following the result.

SUMMARY:
Approximately 40% of members with a positive fecal occult blood result do not continue to followup colonoscopy in Meuhedet. The purpose of this study is to identify the structural, process, carer and patient related causes of undertreatment and suggest appropriate organisational interventions. Using both quantitative and qualitative methods, the investigators will identify organisational and personal barriers to completion of followup of positive FOBT.

DETAILED DESCRIPTION:
Colorectal cancer is the second in incidence and mortality among malignant tumors. Early detection of the disease is an effective means of reducing mortality and is possible through a fecal occult blood test. In the case of a positive result colonoscopy is required. In Israel, about 30% of people with a positive occult blood test do not perform a follow-up test.

The aim of the study is to identify existing barriers to undergoing colonoscopy in a normal-risk population and improving adherence through different intervention mechanisms. At the end of the study we will describe effective intervention models at three levels: the patient, physicians and the organisation to improve early detection of colon cancer.

Innovation of the Study

* It will focus on the normal-risk population groups in Israel with a positive occult blood that didn't undergo colonoscopy.
* Will identify the barriers in diverse populations
* Will review the accessibility of diagnostic facilities forcolon cancer in Israel.
* Will propose intervention programs to improve adherence at all levels in the process.

Study Methods: A prospective study sing both both quantitative and qualitative methods in Meuhedet Health Services Target Population: Health system managers, physicians, and patients (a representative sample of 200 patients adhere colonoscopy and 600 that didn't adhere). Data collection databases from Meuhedet. The study will include questionnaires, focus groups and interviews.

Stages of the study:

1. Describe the magnitude of the problem
2. Map the barriers to adherence with colonoscopy recommendations among patients, physicians and geographic availability of colonoscopies facilities.
3. Suggest intervention models for physicians, patients and organisations according to the information provided by data collection.
4. Recommendation to decision makers on the implementation of national policy intervention.

Data processing: will use SPSS statistical analysis with the types of variables.

ELIGIBILITY:
Inclusion Criteria:

Members of MHC aged 50-74 who completed a fecal occult blood test during the study period.

Exclusion Criteria:

None

Ages: 51 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a representative sample of Meuhedet members who adhered / did not adhere to followup of a positive fecal occult blood test using colonoscopy
Sampling Method: Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Variables related to non-completion of colonoscopy following a positive fecal occult blood test | 18 months
  Quantitative and qualitative variables associated with non-completion of colonoscopical followup among members with a positive screening fecal occult test result: Availability and distance variables (hours, kms), Patient knowledge and awareness (questionnaire scores), Physician knowledge and awareness (qualitative data),

CONTACTS AND LOCATIONS:
Overall Officials: Revital Azulay, MSC, Principal Investigator — Meuhedet Health Care
Locations (1):
- Meuhedet, Tel Aviv, Israel

REFERENCES:
- [Derived] Azulay R, Valinsky L, Hershkowitz F, Magnezi R. Is the patient activation measure associated with adherence to colonoscopy after a positive fecal occult blood test result? Isr J Health Policy Res. 2018 Dec 21;7(1):74. doi: 10.1186/s13584-018-0270-8. PMID 30577883